CLINICAL TRIAL: NCT03714620
Title: A Randomized, Controlled Trial of Intravenous Sub-dissociative Ketamine at Two Doses for Analgesia in the Emergency Department
Brief Title: Sub-dissociative Dose Ketamine Dosing Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Shannon Lovett, Associate Professor of Department of Emergency Medicine, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 211328
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: The sequence will be generated using randomization permuted blocks of 2 and 4 patients, with the allocated dose revealed using an online randomization module within the REDCap data management system.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study investigators, patients and clinicians except the clinical pharmacist will be blinded to the study treatment allocation. Treatment will be prepared and blinded by the ED clinical pharmacist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 0.15 mg/kg IV Ketamine (Active Comparator)
  Interventions: Drug: Ketamine
- 0.3 mg/kg IV Ketamine (Active Comparator)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Ketamine 0.15 mg/kg vs. 0.3 mg/kg IVPB over 15 minutes

SUMMARY:
Goal is to determine if in adults presenting to the Emergency Department (ED) with moderate to severe acute pain, Ketamine administered at 0.15 mg/kg will provide similar pain relief to Ketamine administered at 0.3 mg/kg, with fewer adverse effects.

DETAILED DESCRIPTION:
Study investigators will enroll participants who present to the Emergency Department (ED) with moderate to severe acute pain, and require intravenous pain medication. Participants will be double-blinded and randomized to one of the two treatment groups.

Investigators aim to determine if ketamine 0.15 mg/kg IVPB is non-inferior to ketamine 0.3 mg/kg IVBP for the treatment of acute moderate to severe pain in the Emergency Department (ED). Study investigators hypothesize that in adults presenting to the ED with moderate to severe acute pain, SDK administered at 0.15 mg/kg will provide similar pain relief to SDK at 0.3 mg/kg, with reduced adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-59
* Weight 45 - 115 kg
* Acute abdominal, flank, back, musculoskeletal pain, or a headache
* Onset of pain within 7 days
* Pain score of 5 or more
* Requiring intravenous analgesia
* Hasn't been enrolled in this study previously

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Altered mental status rendering the patient unable to consent to the study
* Allergy to ketamine
* Unstable vital signs (systolic blood pressure <90 or >180 mm Hg, pulse rate <50 or >150 beats/minute, and respiration rate <10 or >30 breaths/minute)
* History of acute head or eye injury, seizure, intracranial hypertension
* Chronic pain
* Renal or hepatic insufficiency
* Known alcohol or drug use disorder
* Currently under influence of alcohol/opiates
* Acute psychiatric illness

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Lovett, MD, Principal Investigator — Loyola University Chicago, LUMC
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Group: 0.15 mg/kg dose of intravenous ketamine
- High Dose Group: 0.3 mg/kg dose of intravenous ketamine
Period: Overall Study
Arm/Group | Low Dose Group | High Dose Group
Started | 49 | 49
Completed | 49 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.15 mg/kg IV Ketamine | 0.3 mg/kg IV Ketamine | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 39 [36 to 42] | 37 [34 to 41] | 38 [34 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 57
  Male | 19 | 22 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 15 | 13 | 28
  Race: White | 18 | 28 | 46
  Race: Other | 16 | 8 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 49 | 98
Co-morbidities [Number; unit: participants]
  Diabetes | 13 | 3 | 16
  Hypertension | 13 | 8 | 21
  Cancer | 1 | 1 | 2
  Anxiety | 1 | 7 | 8
  Heart Failure | 2 | 1 | 3
  Depression | 3 | 10 | 13
  Obesity | 11 | 9 | 20
Weight [Mean (Inter-Quartile Range); unit: kilograms] | 85 [81 to 90] | 84 [80 to 89] | 84 [80 to 90]
Type of Pain [Count of Participants; unit: Participants]
  Flank | 6 | 4 | 10
  Back | 4 | 2 | 6
  Musculoskeletal | 14 | 16 | 30
  Headache | 2 | 4 | 6
  Abdominal | 23 | 23 | 46
Duration of Pain [Count of Participants; unit: Participants]
  <24 hours | 21 | 28 | 49
  2 days | 9 | 9 | 18
  3-7 days | 19 | 12 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score From Baseline to 30 Minutes Post Initiation of Drug Administration
Description: Change in numerical pain score (NRS) from time 0 to time 30 min. The NRS ranges from 0 to 10 with higher scores indicating more pain.
Time Frame: 30 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 0.15 mg/kg IV Ketamine | 0.3 mg/kg IV Ketamine
Number analyzed (Participants) | 49 | 49
score on a scale | 3.8 [3.0 to 4.7] | 3.5 [2.7 to 4.3]

2. Secondary Outcome: Change in Pain Score From Baseline to 15 Minutes
Description: Change in numerical pain score (NRS) from time 0 to time 15 min. The NRS ranges from 0 to 10 with higher scores indicating more pain.
Time Frame: 15 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 0.15 mg/kg IV Ketamine | 0.3 mg/kg IV Ketamine
Number analyzed (Participants) | 49 | 48
score on a scale | 3.6 [2.7 to 4.4] | 4.8 [4.0 to 5.6]

3. Secondary Outcome: Change in Pain Score From Baseline to 60 Minutes
Description: Change in numerical pain score (NRS) from time 0 to time 60 min. The NRS ranges from 0 to 10 with higher scores indicating more pain.
Time Frame: 60 minutes
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 0.15 mg/kg IV Ketamine | 0.3 mg/kg IV Ketamine
Number analyzed (Participants) | 49 | 49
score on a scale | 3.7 [2.9 to 4.6] | 3.5 [2.6 to 4.4]

4. Secondary Outcome: Number of Participants Who Need Additional Pain Medication at 30 Minutes
Description: Patient request for additional pain medications at 30 minutes post initiation of drug administration
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 0.15 mg/kg IV Ketamine | 0.3 mg/kg IV Ketamine
Number analyzed (Participants) | 49 | 49
Participants | 1 | 0

5. Secondary Outcome: Number of Patients Who Need Rescue Medications at 60 Minutes
Description: Patient request for additional pain medications at 60 minutes
Time Frame: 60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 0.15 mg/kg IV Ketamine | 0.3 mg/kg IV Ketamine
Number analyzed (Participants) | 49 | 49
Participants | 2 | 4

6. Secondary Outcome: Adverse Effects at 30 Min
Description: Patients were asked if they had any adverse effects at 30 minutes including nausea, dizziness, headache, hallucinations, etc.
Time Frame: 30 minutes
Measure: Number; unit: participants
Arm/Group | 0.15 mg/kg IV Ketamine | 0.3 mg/kg IV Ketamine
Number analyzed (Participants) | 49 | 49
participants
  Fatigue | 18 | 20
  Dizziness | 21 | 16
  Headache | 16 | 11
  Feeling of Unreality | 8 | 6
  Hearing Changes | 0 | 2
  Vision Changes | 4 | 6
  Mood Alteration | 4 | 6
  Discomfort | 15 | 21
  Hallucinations | 2 | 3

ADVERSE EVENTS:
Time Frame: 60 minutes
Description: The reported adverse "effects" were considered known and anticipated with this drug regimen so very much anticipated and many very mild.
Arm/Group | 0.15 mg/kg IV Ketamine | 0.3 mg/kg IV Ketamine
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 28/49 | 31/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.15 mg/kg IV Ketamine (N=49) | 0.3 mg/kg IV Ketamine (N=49)
Fatigue (General disorders) | 18 (18) | 20 (20) — Experienced feeling of fatigue
Dizziness (Nervous system disorders) | 21 (21) | 16 (16) — Feeling dizzy
Headache (General disorders) | 16 (16) | 11 (11) — Feeling Headache
Feeling of Unreality (General disorders) | 8 (8) | 6 (6) — Feeling out of body/unreality
Hearing Changes (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Vision Changes (Eye disorders) | 4 (4) | 6 (6)
Mood Alteration (Psychiatric disorders) | 4 (4) | 6 (6)
Discomfort (General disorders) | 16 (16) | 21 (21)
Hallucinations (Psychiatric disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT03714620/Prot_SAP_000.pdf